CLINICAL TRIAL: NCT02184845
Title: Open, Prospective, Single Cohort, Multi-centre Study Evaluating the NobelActive 3 mm Implant Immediately Restored With Single Crowns in the Maxillary Lateral Incisor Area or Mandibular Central or Lateral Incisor Area
Brief Title: A 5 Year Clinical Study on NobelActive 3 mm Implants
Acronym: NA 3 MM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T 176
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2020-11

CONDITIONS: Single Tooth Implant
Keywords: single tooth implant; supported restoration(s); maxillary lateral incisor; mandibular central incisor; lateral incisor; areas of the mouth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- NobelActive 3.0 (Experimental)
  Interventions: Device: Implant NobelActive 3.0

INTERVENTIONS:
Device: Implant NobelActive 3.0

SUMMARY:
Multi-centre study evaluating the NobelActive 3.0 mm implant immediately restored with single crowns in the maxillary lateral incisor area or mandibular central or lateral incisor area.

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent from the subject.
* The subject shall be at least 18 years of age and have passed secession of growth.
* The subject shall be in need of one or more single tooth implant supported restoration(s) in the maxillary lateral incisor or mandibular central or lateral incisor areas of the mouth.
* The subject shall have natural tooth roots present on both sides adjacent to the implant position.
* The subject must be in such a physical and mental condition that a 5-year follow-up period can be carried out without foreseeable problems.
* The subject shall have sufficient bone volume at the implant site for placing a NobelActive 3.0 mm implant with a length of at least 10 mm.
* The subject as well as the implant site shall fulfill criteria for immediate provisionalization within 24 hours. A minimum insertion torque of 35 Ncm without further rotation is required.
* The implant site shall be free from tooth remnants.
* If the implant is placed in an extraction site, the extraction socket should have at least 3 intact walls. A dehiscence defect of up to 3 mm is permitted on the fourth wall.
* If the implant is placed in an extraction site, proper and thorough debridement of the extraction socket should be performed.
* The subject shall be healthy and compliant with good oral hygiene.
* The subject shall have a favorable and stable occlusal relationship.

Exclusion Criteria:

* The subject is not able to give her/his informed consent of participating
* Health conditions, which do not permit the surgical treatment.
* Reason to believe that the treatment might have a negative effect on the subject's total situation (psychiatric problems), as noted in subject records or in subject history.
* Any disorders in the planned implant area such as previous tumours, chronic bone disease or previous irradiation.
* Teeth in positions adjacent to the implant site with ongoing infections, endodontic or peri-odontal problems.
* Alcohol or drug abuse as noted in subject records or in subject history.
* Heavy smoking (>10 cigarettes/day).
* Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake.
* Any other disease or medication that might have an influence on the involved tissues, such as intake of bisphosphonates, treatment with heparine, osteogenesis imperfecta, osteoporosis etc.
* Severe bruxism or other destructive habits.
* If the implant is not able to withstand a final torque of 35 Ncm without further rotation, or if the implant for any other reason cannot be immediately provisionalized, as judged by the clinician, the implant will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-01; Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Marginal bone level changes | 5 years
  Marginal bone level changes over time around the NobelActive 3.0 mm implant

REFERENCES:
- [Derived] Weigl P, Trimpou G, Hess P, Kolinski M, Bellucci G, Trisciuoglio D, Friberg B, Leziy S, Al-Nawas B, Wagner W, Pozzi A, Ottria L, Wiltfang J, Behrens E, Vasak C, Zechner W. Esthetically driven immediate provisionalization in the anterior zone: 5-year results from a prospective study evaluating 3.0-mm-diameter tapered implants. Clin Oral Investig. 2024 Jul 31;28(8):460. doi: 10.1007/s00784-024-05832-x. PMID 39083185